CLINICAL TRIAL: NCT06623552
Title: Relationship Between Cervical Pain and Temporomandibular Dysfunction Craniovertebral Angle, Jaw Functional Limitation and Cervical Mobility
Acronym: TMJ
Status: Completed | Type: Observational
Sponsor: Yeditepe University (Other)
Responsible Party: Sponsor
Other Study IDs: TMJ
Record Dates: First submitted 2024-09-30; First posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Temporomandibular Disorder
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control Group: the population without cervical pain or with a cut off value of less than 15 for neck pain and disability score(NPDS) were selected as the control group
  Interventions: Other: Neck Pain and Disability Scale (NPDS); Other: Fonseca Anamnestic Index (FAI); Other: Evaluation of Jaw Functional Limitation
- Study Group: the population without cervical pain or with a cut off value of more than 15 for neck pain and disability score(NPDS) were selected as the study group
  Interventions: Other: Neck Pain and Disability Scale (NPDS); Other: Fonseca Anamnestic Index (FAI); Other: Evaluation of Jaw Functional Limitation

INTERVENTIONS:
Other: Neck Pain and Disability Scale (NPDS) — The Turkish version of the Neck Pain and Disability Scale (NPDS), developed by Wheeler et al., was used for individuals with neck pain. The severity of neck pain is evaluated on a 5-point Likert scale; where 0 indicates "no pain" and 4 indicates "very severe pain". The score is higher in those with upper extremity symptoms.The cut-off value of this scale was set to 15 to detect disability-related neck pain.The cut-off value is mandatory to evaluate a patient or a particular group of patients for clinically significant neck pain by distinguishing it from insignificant pain
Other: Fonseca Anamnestic Index (FAI) — It is a questionnaire consisting of 10 questions, including pain during the period, parafunctional habits, movement restriction, clicking, malocclusion, emotional stress.In this study, clinical signs relevant to each severity category of Fonseca's anamnestic index were used to detect the frequency of symptoms and to characterize the symptoms and clinical findings of TMD.The Turkish version of Fonseca's Anamnestic Index (FAI) questionnaire was used to assess the symptom severity.
Other: Evaluation of Jaw Functional Limitation — The Jaw Functional Limitation Scale (JFLS) was developed as an 8-item scale for general functional limitation in the jaw. In the light of the obtained items and supporting psychometric data, it has been expanded and re-developed to include the verbal and non-verbal communication limitations that occur in a 20-item tool16 JFLS-20 is a tool with three structure contents (chewing, vertical mobility of jaw state and emotional and verbal statement) to evaluate functional state.Difficulty performing a determined task is graded from 0 (without limitation) to 10 (severe limitation). Higher scores are a more serious sign of functional limitation.

SUMMARY:
The aim of this study is to examine temporomandibular dysfunctions, jaw functional limitation, cervical mobility and craniovertebral angles and possible relations between individuals with cervical pain and individuals without cervical pain and to compare the this four variables between the two groups.

DETAILED DESCRIPTION:
This study was conducted with 129 individuals (mean age 34.08:years, M/F=52/77) to determine the possible relationships between Cervical Pain and Temporomandibular Dysfunction, Craniovertebral Angle, Jaw Functional Limitation and Cervical Mobility. Pati,ents were assessed with Neck Pain and Disability Questionnaire , Fonseka Anamnestic Index , goniometric measurements, ,Cervical Mobility Measurement. JFSL-20 questionnaire and Craniovertebral Angle measurement was made by photographic method.

ELIGIBILITY:
Inclusion Criteria:

Neck pain disability score below 15 Not having painting problem for TME Being in the age range of 18-50 Volunteering to participate in the study

Exclusion Criteria:

* he presence of any orthopedic and / or neurological problem that may prevent evaluations.

Being diagnosed with any psychiatric disorder Situations that will prevent evaluation or communication

* Illiterate individuals
* Head, neck and maxillofacial surgery operation history
* Conditions in systemic pathological conditions such as malignant condition, fracture and rheumatoid arthritis

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All individuals in the study were included on a voluntary basis.All participants were informed about the study before the evaluations and the consent form was signed (Appendix- ).All necessary evaluations for the study were carried out on the same day.During the study, both the participants in the study group and the participants in the control group completed the evaluation completely.No health problems were observed in any participant during and after the evaluations.
Sampling Method: Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Neck Pain and Disability Scale (NPDS): | one day

SECONDARY OUTCOMES:
Fonseca Anamnestic Index (FAI): | one day

CONTACTS AND LOCATIONS:
Locations (1):
- Yeditepe University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided